CLINICAL TRIAL: NCT00891891
Title: Psychosocial Adjustment of Adolescents With Spina Bifida
Acronym: CHATS
Status: Active, not recruiting | Type: Observational
Sponsor: Loyola University Chicago (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Grayson N. Holmbeck, PhD, Principal Investigator, Loyola University Chicago
Other Study IDs: R01NR016235 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Spina Bifida
Keywords: spina bifida; psychosocial adjustment; adolescence; emerging adulthood
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spina Bifida: 140 children with spina bifida (ages 8-15)

SUMMARY:
The purpose of this longitudinal study is to evaluate a developmentally-oriented bio-neuropsychological model of adjustment in youth and young adults with spina bifida. The theoretical framework for the study is a developmentally-oriented bio-neuropsychosocial model of psychological adjustment.

DETAILED DESCRIPTION:
The purpose of this longitudinal study is to evaluate a developmentally-oriented bio-neuropsychological model of adjustment in youth and young adults with spina bifida (SB). The theoretical framework for the study is a developmentally-oriented bio-neuropsychosocial model of psychological adjustment. Extensive multi-source (i.e., youth, peers, parents, teachers, health professionals, and medical chart) and multi-method (i.e., questionnaires, interviews, neuropsychological testing, and observational) data are collected across several predictor variable domains: (1) biological (i.e., severity of disability, current and past health status, pubertal development), (2) neuropsychological (i.e., executive functions and attention, language pragmatics and inference making skills, emotion recognition), and (3) social (i.e., observed and perceived social behaviors with peers and family). A multidimensional perspective on adjustment will is adopted insofar as the following constructs are assessed: internalizing symptoms (e.g., depression), externalizing symptoms (e.g., aggression), social adjustment, romantic relationship involvement, quality of life and functional status, school performance, vocational achievements, autonomy development, independent living, medical adherence, and the transition to adult medical care. Within the context of this model, several mediation and moderation models are being tested to identify underlying mechanisms for associations between variables and to determine whether variables within one domain can compensate for deficits in another domain.

This longitudinal study of youth with SB includes the following innovations: (1) videotaped social interactions between youth with SB and their close friends, (2) a comprehensive assessment of socially-relevant neuropsychological factors, (3) an extensive multi-respondent questionnaire- and interview-based evaluation of the targets' social adjustment, (4) an interview-based evaluation of the transition to emerging adulthood, and (5) an oversampling of Hispanic families.

Currently, the investigators are collecting Times 4, 5 and 6 longitudinal data on a cohort of 140 youth with SB (ages 8-15 at Time 1, ages 10-17 at Time 2, ages 12-19 at Time 3, ages 14-21 at Time 4, ages 16-23 at Time 5, ages 18-25 at Time 6). Parents and a close friend participate when youth participants are under 18 years of age; when participants are 18 years and older, they are the sole participator. Data is collected via trained research assistants during home visits.

Because of our efforts to select variables that are modifiable, findings of this study will inform interventions designed to address the social difficulties of youth with SB, interventions that facilitate young adults' full participation in the milestones of young adulthood, and the manuals of care that will be developed by the investigators. Moreover, findings will provide policy-relevant information to improve the transition to adult medical care for individuals with this debilitating birth defect.

ELIGIBILITY:
Inclusion criteria for youth with SB were:

1. a diagnosis of SB (types included myelomeningocele, lipomeningocele, myelocystocele),
2. age 8-15 years at Time 1,
3. ability to speak and read English or Spanish,
4. involvement of at least one primary custodial caregiver,
5. residence within 300 miles of the laboratory (to allow for home visits to collect data).

Latino families were intentionally oversampled to better study this subpopulation of youth with SB, given their prevalence.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with spina bifida (ages 8-15) and their families and close friends
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2005-09; Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Transition to Adult Healthcare Interview and Coding System | when youth are 18 years old; 8-10 years after the start of the study
  Young adults will be asked questions about their pediatric care and whether they have transitioned to a primary care provider and/or an adult-oriented health care service. A quantitative coding system was developed by this team to score each participant on their transition status. The success of the transition is assessed separately for each provider, is based on an assessment of whether or not the youth has experienced transition-related meetings and includes an assessment of each youth's subjective opinion regarding their transition status. Finally, the success of the transition is assessed by examining how they manage health-related complications.
Medical History Questionnaire | when youth are 18 years old; 8-10 years after the start of the study
  Data regarding adherence will be obtained from the Medical History Questionnaire. The Medical History Questionnaire was adapted from the Parent-Report of Medical Adherence in Spina Bifida Scale (PROMASB, Holmbeck et al., 1998), which was developed for a previous study on youth with spina bifida by the same investigator. The measure is designed to obtain disease-specific medical information, including bowel and bladder functioning, ambulation, medications, providers and frequency of medical care, and surgery history.
Spina Bifida Self-Management Profile | when youth are 18 years old; 8-10 years after the start of the study
  The Spina Bifida Self-Management Profile (SBSMP) was developed by Wysocki and Gavin (2006). The SBSMP is a 14-question, structured interview addressing seven dimensions of the spina bifida regimen, including appointment keeping, bowel control program, skin and wound care, exercise, medications, clean intermittent catheterization, and dealing with urinary tract infections. Item content, wording, and scoring was developed with the consultation of medical experts. Internal consistency is acceptable, with an alpha of .66 for mothers of children with spina bifida (Wysocki & Gavin, 2006). In this study, the SBSMP will be administered as a questionnaire rather than in interview format.

SECONDARY OUTCOMES:
Sharing of Spina Bifida Management Responsibilities | when youth are 18 years old; 8-10 years after the start of the study
  A self-report measure of psychosocial adjustment, the Sharing of Spina Bifida Management Responsibilities (SOSBMR) is adapted from the Diabetes Family Responsibility Questionnaire (DFRQ; Anderson, Auslander, Jung, Miller, & Santiago, 1990). The DFRQ consists of 17 items that describe diabetes and general health-related situations or tasks relevant to children and adolescents. Reporters rate each task on a three-point Likert scale as a child, parent, or shared responsibility. Participants were instructed to check the N/A box if the task is not part of their care. Higher scores indicate greater child responsibility. Items fall into three subscales, including general health maintenance, regimen tasks, and social presentation of diabetes.
Spina Bifida Readiness for Self-Management | when youth are 18 years old; 8-10 years after the start of the study
  A self-report measure of psychosocial adjustment, the Spina Bifida Readiness for Self-Management questionnaire is a self-report questionnaire adapted from a model of stages of change relating to smoking cessation (DiClemente et al., 1991). The Spina Bifida Readiness for Self-Management questionnaire instructs respondents to indicate the frequency of behaviors over the prior six months across 14 items relating to appointment keeping, bowel control program, skin and wound care, exercise, medications, clean intermittent catheterization, and dealing with urinary tract infections. The questionnaire also assesses the presence and frequency of spina bifida-related complications (i.e., pressure sores/wounds on skin) over the previous six months, and co-occurring medical disorders (i.e., Type II diabetes).
Spina Bifida Independence Survey | when youth are 18 years old; 8-10 years after the start of the study
  A self-report measure of psychosocial adjustment, the Spina Bifida Independence Survey (SBIS) is adapted from the Diabetes Independence Survey (DIS; Wysocki et al., 1996). The DIS is a brief measure of the parent's evaluation of the child's growth and development of diabetes knowledge and skills among children and adolescents with diabetes. Participants respond "yes" or "no" to whether their child has mastered a disease-related skill (e.g. "Can your child state each type of insulin he/she uses?")
Spina Bifida Barriers to Adherence Questionnaire (SBBAQ) | when youth are 18 years old; 8-10 years after the start of the study
  A self-report measure of psychosocial adjustment, the Spina Bifida Barriers to Adherence Questionnaire (SBBAQ) is a self-report measure assessing multiple spina bifida-related barriers, adapted from the Barriers to Diabetes Adherence (BDA) measure for adolescents (Mulvaney, et al., 2011). The SBBAQ instructs subjects to indicate how true to them different statements are on a five-point likert scale (1 = Completely Not True to 5 = Completely True).
Spina Bifida Self-Efficacy Survey | when youth are 18 years old; 8-10 years after the start of the study
  A self-report measure of psychosocial adjustment, the Spina Bifida Self-Efficacy Survey (SBSS) is a self-report questionnaire adapted from a measure of self-efficacy and self-management for adolescents with diabetes (Iannotti et al., 2006). The SBSS instructs respondents to indicate how sure they are they can complete tasks on their own all of the time across 17 items, on a five-point likert scale (i.e., 1 = Completely Unsure to 5 = Completely Sure).

CONTACTS AND LOCATIONS:
Overall Officials: Grayson N Holmbeck, PhD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: Lab's website — http://chatslab.weebly.com/
- See also: Holmbeck's professional website — http://www.luc.edu/psychology/facultystaff/holmbeck_g.shtml